CLINICAL TRIAL: NCT02970747
Title: A Non-interventional Study of Carfilzomib (Kyprolis®) in Combination With Lenalidomide (Revlimid®) and Dexamethasone or Carfilzomib in Combination With Dexamethasone Alone or Carfilzomib in Combination With Daratumumab (Darzalex®) and Dexamethasone in Patients With Multiple Myeloma Who Have Received at Least One Prior Therapy
Brief Title: Non-interventional Study of Kyprolis® in Combination With Revlimid® and Dexamethasone or Dexamethasone Alone or in Combination With Darzalex® and Dexamethasone in Multiple Myeloma Patients
Acronym: CARO
Status: Completed | Type: Observational
Sponsor: iOMEDICO AG (Industry)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: IOM-070337
Record Dates: First submitted 2016-11-10; First posted 2016-11-22 (Estimated); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Multiple Myeloma in Relapse
MeSH Terms: interventions — carfilzomib

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Car/Len/Dex (KRd): Patients treated with carfilzomib, lenalidomide and dexamethasone dosage form, dosage, frequency and duration of treatment according to current SmPC
  Interventions: Drug: Carfilzomib
- Car/Dex (Kd): Patients treated with carfilzomib and dexamethasone dosage form, dosage, frequency and duration of treatment according to current SmPC
  Interventions: Drug: Carfilzomib
- Car/Dex/Dara (KdD): Patients treated with carfilzomib, dexamethasone and daratumumab dosage form, dosage, frequency and duration of treatment according to current SmPC
  Interventions: Drug: Carfilzomib

INTERVENTIONS:
Drug: Carfilzomib — In accordance with SmPC.
  Other Names: Kyprolis®

SUMMARY:
The objective of this non-interventional study (NIS) is to evaluate patients' adherence and persistence to carfilzomib therapy in combination with lenalidomide and dexamethasone or in combination with dexamethasone alone or in combination with daratumumab and dexamethasone in adult patients with multiple myeloma (MM) who have received at least one prior therapy in a real-life setting.

DETAILED DESCRIPTION:
The dual combination of lenalidomide (Revlimid®) (R) and dexamethasone (d) (Rd) as well as the dual combination of bortezomib (Velcade®, V) and dexamethasone (Vd) are standard regimens to treat MM patients who have received at least one prior therapy. Recently published clinical data indicate that the next-generation proteasome inhibitor carfilzomib (Kyprolis®) (K) may substantially change the treatment paradigm for patients with relapsed or refractory MM (RRMM).1 Three pivotal trials were conducted leading to market authorization of carfilzomib in combination with lenalidomide and dexamethasone or in combination with dexamethasone alone or in combination with dexamethasone and daratumumab for the treatment of MM patients who have received at least one prior therapy.

ASPIRE, NCT010803912 To compare the efficacy and safety of carfilzomib in combination with Rd (KRd) with the dual combination therapy Rd, a randomized, multicenter, open-label phase III study was performed in patients with relapsed MM (RMM). After cycle 18, carfilzomib was discontinued in the KRd arm, but Rd administration was continued thereafter until disease progression. The trial met its primary endpoint progression-free survival (PFS) (Hazard Ratio (HR) for progression or death, 0.69; p=0.0001). Median PFS was 26.3 months with KRd treatment compared to 17.6 months with Rd treatment. The study further demonstrates that carfilzomib improves patients' overall survival (OS) rate at 24 months (KRd, 73.3% vs. Rd, 65.0%; HR for death, 0.79; p=0.04) and overall response rate (ORR) (KRd, 87.1% vs. Rd, 66.7%; p<0.001). Objective assessment of adverse events (AEs) and patient-reported outcomes (PRO) revealed that the benefit-risk ratio is favorable for the three-drug combination KRd.

ENDEAVOR, NCT015688663 To compare the efficacy and safety of the dual combination therapy Kd with the dual combination therapy Vd, a randomized, multicenter, open-label phase III study was performed in patients with RRMM. Patients in both arms received treatment until progression. Results of the preplanned interim analysis show, that the trial met its primary endpoint PFS (HR for progression or death, 0.53; p<0.0001). Median PFS was 18.7 months with Kd treatment compared to 9.4 months with Vd treatment. In addition, the Kd combination therapy demonstrated superiority over the Vd combination therapy for secondary objectives, like ORR (77% vs. 63%; p<0.0001) and median duration of response (DOR) (21.3 months vs. 10.4 months). OS data were not available at time of analysis. Despite higher rates for cardiac and renal failure as well as higher incidence of hypertension and dyspnea in the Kd arm, carfilzomib given as a 30 min infusion has an acceptable safety profile, particularly with respect to lower peripheral neuropathy events. The number of patients who had ≥ grade 2 peripheral neuropathy was significantly higher in the Vd group than in the Kd group (32% vs. 6%). In conclusion, data of the ENDEAVOR study demonstrate, that carfilzomib given in combination with dexamethasone has a favorable benefit-risk profile and provides an important new treatment option for patients with RRMM.

CANDOR, NCT031586884-7 To compare the efficacy and safety of carfilzomib in combination with dexamethasone and daratumumab (KdD) with the dual combination therapy Kd, a randomized, multicenter, open-label phase III study was performed in patients with RRMM. Patients in both arms received treatment until progression. The trial met its primary endpoint PFS (HR for progression or death, 0.59). Median PFS was 28.6 months in the KdD arm and 15.2 months with Kd treatment with a median follow-up time of 27.8 months and 27.0 months, respectively. Further, KdD treatment demonstrates improved response rates by providing deeper responses. ORR was 84% (with 29% complete response (CR) or better) for KdD treatment and 75% (with 10% CR or better) for Kd treatment (p=0.0080). The minimal residual disease (MRD) negative CR rate at 12 months is nearly 10-times higher with KdD (12.5%) compared to Kd (1.3%). Overall, the safety profile is consistent with the known safety profiles of each agent, with the exception of an imbalance in treatment-emergent fatal AEs, which might be partially explained by longer treatment exposure, age, and frailty status.

Up to now, no real-life data on patients' adherence, persistence, quality of life (QoL) and patterns of use, effectiveness and safety of the KRd,the Kd and the KdD regimen have been systematically collected and analyzed. Thus, after market approval of KRd, Kd and KdD as treatment for patients with MM who have received at least one prior therapy, the purpose of the CARO NIS is to evaluate patients' adherence, persistence and QoL as well as effectiveness and safety of both regimens in a real-life setting.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older.
* Patients with MM who have received at least one prior therapy.
* Indication for treatment as assessed by the treating physician.
* Decision for second- or subsequent-line treatment with the combination therapy carfilzomib/ lenalidomide/ dexamethasone or carfilzomib/ dexamethasone or carfilzomib/ dexamethasone/ daratumumab
* Signed written informed consent.
* Criteria according to the current Summary of Product Characteristics (SmPC) for Kyprolis® (Carfilzomib)

Exclusion Criteria:

* Contraindications according to the current SmPC for Kyprolis® (Carfilzomib)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with multiple myeloma (MM) who have received at least one prior therapy
Sampling Method: Probability Sample
Enrollment: 359 (Actual)
Dates: Start 2016-10-25 (Actual); Primary Completion 2025-04-26 (Actual); Study Completion 2025-04-26 (Actual)

PRIMARY OUTCOMES:
Patients' adherence and persistence to carfilzomib therapy | Duration of Carfilzomib therapy, up to 24 months after last patient in
  Patients' adherence and persistence to carfilzomib therapy

SECONDARY OUTCOMES:
Patients' adherence and persistence to lenalidomide, dexamethasone and daratumumab therapy | Duration of Carfilzomib therapy, up to 24 months after last patient in
  Patients' adherence and persistence to lenalidomide, dexamethasone and daratumumab therapy

OTHER OUTCOMES:
Median Progression-free Survival (PFS) | up to 24 months after last patient in
  Median Progression-free Survival (PFS)
Overall Survival (OS) rate at 24 months | 24 months
  Overall Survival (OS) rate at 24 months
Median Time to Response (TTR) | up to 24 months after last patient in
  Median Time to Response (TTR)
Median Duration of Response (DOR) | up to 24 months after last patient in
  Median Duration of Response (DOR)
Overall Response Rate (ORR) | up to 24 months after last patient in
  ORR is defined as ≥ Very Good Partial Response (VGPR) + Partial Response (PR)
To assess safety and tolerability measured by adverse events as graded by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v.4.03 | Duration of Carfilzomib therapy (+ 30 days), up to 25 months after last patient in
  AE, SAE and ADR are documented in the eCRF and will be used for safety assessment.
To assess health-related QoL using the validated BOMET-QoL-10 questionnaire | Baseline, 6, 12, 18, 24, End of Treatment (latest up to 24 months after last patient in)
  QoL data will be collected at baseline, after 6, 12, 18, 24 months (during treatment) and at the end of Carfilzomib therapy

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Knauf, Professor, Principal Investigator — Centrum für Hämatologie und Onkologie Bethanien, Germany, 60389 Frankfurt a.M.
Locations (1):
- Centrum für Hämatologie und Onkologie Bethanien, Frankfurt, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Engelhardt M, Ihorst G, Singh M, Rieth A, Saba G, Pellan M, Lebioda A. Real-World Evaluation of Health-Related Quality of Life in Patients With Multiple Myeloma From Germany. Clin Lymphoma Myeloma Leuk. 2021 Feb;21(2):e160-e175. doi: 10.1016/j.clml.2020.10.002. Epub 2020 Oct 24. PMID 33218965